CLINICAL TRIAL: NCT01475149
Title: Effect of Hydroxychloroquine on the Annexin A5 Resistance Assay in Antiphospholipid Antibody-Positive Patients With and Without Systemic Lupus Erythematosus
Brief Title: Effect of HCQ on AnxA5 Resistance Assay in Antiphospholipid (aPL) Positive Patients With and Without Systemic Lupus Erythematosus (SLE)
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 10130
Record Dates: First submitted 2011-11-14; First posted 2011-11-21 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Antiphospholipid Syndrome; Thrombophilia Due to Antiphospholipid Antibody; Systemic Lupus Erythematosus
Keywords: Antiphospholipid syndrome; Antiphospholipid antibodies; Systemic lupus erythematosus; Annexin A5 and Annexin A5 resistance assay
MeSH Terms: conditions — Antiphospholipid Syndrome; Lupus Erythematosus, Systemic | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- aPL positive - group 1: aPL positive with APS, receiving HCQ
  Interventions: Other: Phlebotomy
- aPL positive - group 2: aPL positive with APS and SLE, receiving HCQ
  Interventions: Other: Phlebotomy
- aPL positive - group 3: aPL positive without APS but with SLE, receiving HCQ
  Interventions: Other: Phlebotomy
- aPL positive - group 4: aPL positive without APS or SLE, receiving HCQ
  Interventions: Other: Phlebotomy
- aPL negative - group 1: aPL negative with SLE, receiving HCQ
  Interventions: Other: Phlebotomy
- aPL negative - group 2: aPL negative with SLE, not receiving HCQ
  Interventions: Other: Phlebotomy

INTERVENTIONS:
Other: Phlebotomy — Subjects will have blood drawn at each of the 3 study visits.

SUMMARY:
This 12 week study will observe patients with and without systemic lupus erythematosus who have persistent antiphospholipid antibodies in the blood who are starting a medicine called hydroxychloroquine. It will measure if these patients have a change in a blood test called the annexin A5 resistance assay over that 12 week period.

DETAILED DESCRIPTION:
Antiphospholipid Syndrome (APS) is an autoimmune disorder of blood clotting and pregnancy loss. It is associated with proteins called antiphospholipid antibodies (aPL) in the blood. Blood clotting in this disease occurs for several reasons; one reason involves the interaction of aPL with another protein found on the surface of the cells that line blood vessels (endothelial cells). This protein, called annexin A5 (AnxA5), forms a shield over the surface of these cells. The AnxA5 Resistance Assay is a blood test that can detect when there is a problem with the protective AnxA5 shield on endothelial cell surfaces.

This 12 week study will observe patients with persistent aPL in the blood who are starting a medicine called hydroxychloroquine (HCQ). The primary goal of the study is to compare results of the AnxA5 resistance assay from patients before they start taking HCQ and after they have taken it for 12 weeks to see if the results of the blood test change. Our secondary goal is to measure a variety of other blood tests before and after patients have started taking HCQ; these tests include D-dimer, Activated Protein C (APC) Resistance, and aPL titers/status (LA test, aCL ELISA, aß2GPI ELISA, and anti-Domain-I ß2GPI ELISA).

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65
* new HCQ (200-400 mg/day) treatment (for all but 5 of 10 control subjects - see below)
* persistently positive aPL

Selected Exclusion Criteria:

* Steroid use greater than or equal to the equivalent of prednisone 0.5 mg/kg/day at the time of enrollment
* Heparin use at the time of enrollment
* Any immunosuppressive drug use within 3 months prior to screening
* HCQ use within the past 6 months prior to screening visit
* Another antimalarial agent treatment,
* Pregnant women, minors, mentally disabled, prisoners
* Acute thrombosis within 2 weeks prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For aPL positive groups, subjects must have persistently positive (over at least 12 weeks) antiphospholipid antibodies in the blood.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Annexin A5 resistance assay | 12 weeks
  The primary goal of the study is to compare results of the AnxA5 resistance assay from patients before they start taking HCQ and after they have taken it for 12 weeks to see if the results of the blood test change.

SECONDARY OUTCOMES:
Change in D-dimer | Baseline and 12 weeks
Change in activated protein C (APC) resistance coagulation assay | Baseline and 12 weeks
Change in LA functional coagulation assay | Baseline and 12 weeks
Change in anticardiolipin (aCL) ELISA | Baseline and 12 weeks
Change in anti-B2-glycoprotein-I (aB2GPI) ELISA | Baseline and 12 weeks
Change in anti-Domain-I B2GPI ELISA | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doruk Erkan, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No